CLINICAL TRIAL: NCT01043354
Title: TACTICS (Targeting Adherence to Cholesterol-lowering Therapy to Improve Control Study)
Acronym: TACTICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Narrows Institute for Biomedical Research (Other)
Responsible Party: Principal Investigator, Sundar Natarajan, Attending Physician, Narrows Institute for Biomedical Research
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ADA 7-08-CR-68
Record Dates: First submitted 2010-01-05; First posted 2010-01-06 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-04

CONDITIONS: Hypercholesterolemia
Keywords: cholesterol; diabetes; adherence
MeSH Terms: conditions — Hypercholesterolemia; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- stage-matched intervention (Experimental): Transtheoretical Model-based stage-matched intervention
  Interventions: Behavioral: stage-matched intervention
- framing effects intervention (Experimental): counseling based on prospect theory
  Interventions: Behavioral: framing effects intervention
- attention placebo intervention (Active Comparator): counseling about general health topics
  Interventions: Behavioral: attention placebo intervention

INTERVENTIONS:
Behavioral: stage-matched intervention — 6 monthly tailored telephone-delivered counseling sessions of transtheoretical model-based counseling
  Arms: stage-matched intervention
Behavioral: framing effects intervention — 6 monthly telephone-delivered counseling sessions based on prospect theory
  Arms: framing effects intervention
Behavioral: attention placebo intervention — 6 monthly counseling sessions about general health topics
  Arms: attention placebo intervention

SUMMARY:
Background:

This is a randomized controlled trial (RCT) of two novel behavioral interventions to enhance treatment adherence and improve low-density lipoprotein cholesterol (LDL) in diabetes. Among adults with diabetes, high LDL greatly increases their risk for cardiovascular disease (CVD). Despite the proven efficacy of LDL control(<100 mg/dL) in preventing CVD, the control rate is low. Poor adherence to treatment(diet, exercise and medication) is the main reason for this poor control.

Aims: This study will test two telephone-delivered interventions, a Transtheoretical stage-matched intervention (SMI) and a Prospect theory-based framing effects intervention (FEI). The investigators hypothesize that both SMI and FEI will be more effective in improving LDL control than an attention placebo intervention (API) at 6 months. SMI and FEI will also be more effective in increasing adherence to medications, diet and exercise than API at 6 months.

Methods:

The investigators will recruit 246 adults with diabetes and high LDL despite being on medications. Key outcomes are adherence to diet, exercise and medication, and LDL control. The interventions will be standardized and fidelity of intervention maintained. Using a blinded RCT the investigators will test the effect of SMI and FEI compared to API on LDL control and adherence. All analyses will be intent to treat.

Significance:

This project will provide important information to improve diabetes-related behavior and lead to the implementation of novel interventions for lowering LDL in primary care settings among adults with diabetes. It may also provide the scientific rationale to use such approaches to control other risk factors in diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Adults with diabetes
* LDL greater than or equal to 100
* Cholesterol-lowering drug therapy for > 6 months
* A working telephone
* At least 2 primary care visits in the past 1.5 years

Exclusion Criteria:

* Poor short-term survival (< 1 year)
* Inability to understand English
* Recent major surgery (< 3 months)
* Patients temporarily in the area
* Inability to provide consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2008-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
LDL control | 6 months
medication adherence | 6 months

SECONDARY OUTCOMES:
diet adherence | 6 months
exercise adherence | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sundar Natarajan, MD, M.Sc., Principal Investigator — VA New York Harbor Healthcare System
Locations (1):
- VA New York Harbor Healthcare System, NY and BK Campuses, New York, New York, United States